CLINICAL TRIAL: NCT06998160
Title: Changsha Stomatological Hospital
Brief Title: Analysis of the Factors Influencing the Occurrence of Peri-implant Inflammation in Patients With Oral Implant Repair and Study on the Maintenance Effect of Subgingival Sandblasting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hui Xie (Other Government)
Responsible Party: Sponsor-Investigator, Hui Xie, Principal Investigator, Changsha Stomatological Hospital
Organization: Changsha Stomatological Hospital (Other Government)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: No. 2023-023
Record Dates: First submitted 2025-04-24; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-04

CONDITIONS: Peri-implantitis; Dental Implant Complications; Periodontal Inflammation; Gingival Diseases
MeSH Terms: conditions — Peri-Implantitis; Gingival Diseases | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): The control group was given ultrasonic subgingival curettage. With Swiss EMS ultrasonic therapy instrument, both the operator and the patient should wear safety goggles before operation. After the operator guides the patient to gargle, the mouth opener should be placed to perform ultrasonic subgingival curetting. The debridement time of the implant area should be controlled within 6 minutes, and the debridement time of other sites should be 5 s.
  Interventions: Other: control group
- glycine subgingival sandblasting group and erythritol subgingival sandblasting group (Other): Given glycine subgingival sandblasting group glycine subgingival sandblasting group. Swiss EMS ultrasonic therapy instrument and EMS glycine sandblasting were used. Before the operation, both parties should wear safety glasses and place the mouth opener after the patient gargled. The location of sandblasting was selected to be 1-2 mm below the gingiva. During the operation, the time of sandblasting in the planting area should be controlled within 10 minutes, and then the time of sandblasting at other sites with the same amount of water and power should be controlled within 5s. After sandblasting, the patient's mouth was continuously rinsed with normal saline for 20s. After the operation, the patient was informed of the precautions after the operation, and the patient was instructed to master the correct oral maintenance method, pay attention to maintaining the cleanliness around the implant, and adhere to regular periodontal maintenance.
  Interventions: Other: glycine subgingival sandblasting group and erythritol subgingival sandblasting group

INTERVENTIONS:
Other: glycine subgingival sandblasting group and erythritol subgingival sandblasting group — Given glycine subgingival sandblasting group glycine subgingival sandblasting group. Swiss EMS ultrasonic therapy instrument and EMS glycine sandblasting were used. Before the operation, both parties should wear safety glasses and place the mouth opener after the patient gargled. The location of sandblasting was selected to be 1-2 mm below the gingiva. During the operation, the time of sandblasting in the planting area should be controlled within 10 minutes, and then the time of sandblasting at other sites with the same amount of water and power should be controlled within 5s. After sandblasting, the patient's mouth was continuously rinsed with normal saline for 20s. After the operation, the patient was informed of the precautions after the operation, and the patient was instructed to master the correct oral maintenance method, pay attention to maintaining the cleanliness around the implant, and adhere to regular periodontal maintenance.
  Arms: glycine subgingival sandblasting group and erythritol subgingival sandblasting group
Other: control group — The control group was given ultrasonic subgingival curettage. With Swiss EMS ultrasonic therapy instrument, both the operator and the patient should wear safety goggles before operation. After the operator guides the patient to gargle, the mouth opener should be placed to perform ultrasonic subgingival curetting. The debridement time of the implant area should be controlled within 6 minutes, and the debridement time of other sites should be 5 s.
  Arms: control group

SUMMARY:
Abstract Objective The purpose of this study was to analyze the factors affecting the occurrence of peri-implant inflammation in patients with oral implant repair, and to explore the effect of subgingival sandblasting technology on the maintenance of microecology around the implant, so as to provide a basis for optimizing clinical prevention and treatment strategies.

Method Ninety-six patients with early periimplantitis treated in our hospital from July 2022 to July 2024 were selected as the inflammation group. All patients were randomly divided into control group, glycine subgingival sandblasting group and erythritol subgingival sandblasting group (n=32). The clinical therapeutic effect of the two groups was compared. A total of 102 patients who underwent oral implant repair in our hospital during the same period without peri-implant inflammation were selected as the group without inflammation. The independent risk factors of peri-implant inflammation were analyzed.

ELIGIBILITY:
Inclusion Criteria Clinical diagnosis of peri-implantitis (PD ≥4 mm with BOP/suppuration)

At least one functional dental implant in place for ≥6 months

Willing and able to maintain standard oral hygiene protocol

No antibiotic or anti-inflammatory drug use in the past 30 days

Absence of uncontrolled systemic diseases (e.g., diabetes, hypertension)

Complete baseline clinical data available (medical history, radiographs, lab results)

Exclusion Criteria Acute oral infections requiring immediate treatment

History of radiation therapy to the head/neck region

Severe uncontrolled periodontal disease

Active malignancy or current cancer treatment

Coagulation disorders or anticoagulant therapy

Pregnancy or lactation

Cognitive impairment affecting compliance

Allergy to glycine or erythritol compounds

Non-Inflammatory Group Additional Criteria Successful implant placement with no signs of inflammation (PD ≤3 mm, no BOP)

Matched to study group by age (±5 years) and implant location

Meets all other inclusion/exclusion criteria regarding systemic health

Note: All participants must provide informed consent. Healthy volunteers without implants are not eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-03-09 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Change in Plaque Index (PLI) Score | Baseline, 3 months, 6 months.
  Change in Plaque Index (PLI; scored 0-3) from baseline to 3 and 6 months post-treatment, comparing subgingival sandblasting (glycine/erythritol) versus standard ultrasonic curettage. Higher scores indicate greater plaque accumulation.
Change in Bleeding Index (BI) Score | Baseline, 3 months, 6 months.
  Change in Bleeding Index (BI; scored 0-3) from baseline to 3 and 6 months post-treatment, comparing interventions. Higher scores indicate more severe gingival bleeding.
Change in Probing Depth (PD) | Baseline, 3 months, 6 months.
  Change in Probing Depth (PD; measured in millimeters) from baseline to 3 and 6 months post-treatment, comparing interventions. Deeper pockets indicate worse peri-implant inflammation.

SECONDARY OUTCOMES:
Inflammatory Biomarker Levels (IL-6, IL-1β) | Baseline, 1 month post-treatment, 3 months post-treatment, 6 months post-treatment
  Change in pro-inflammatory cytokine levels measured in peri-implant crevicular fluid via ELISA across treatment groups.

OTHER OUTCOMES:
Peri-Implantitis Recurrence Rate | 12 months post-treatment
  Incidence of peri-implant inflammation recurrence (PD ≥5mm with bleeding/suppuration) in treated patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Changsha Stomatological Hospital, Changsha, China